CLINICAL TRIAL: NCT03573076
Title: Treatment of Photodamaged Skin of the décolleté With Fractional Laser, Radio-frequency Microneedling, and Photodynamic Therapy
Brief Title: Treatment of Photodamaged Skin of the décolleté
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The second study arm including radio-frequency microneedling was withdrawn due to availability of newer treatment options.
Sponsor: Merete Haedersdal (Other)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Professor, Physician Consultant, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-000189-12
Record Dates: First submitted 2018-06-06; First posted 2018-06-29 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Photodamaged Skin
MeSH Terms: interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Thulium laser + photodynamic therapy (Experimental): Non-ablative Thulium laser (NAFL) + Photodynamic therapy combination treatment
  Interventions: Combination Product: Photodynamic therapy; Device: Non-ablative Thulium laser (NAFL)
- RF microneedles + photodynamic therapy (Experimental): Radio-frequency microneedles (RF-MN) + Photodynamic therapy combination treatment
  Interventions: Combination Product: Photodynamic therapy; Device: Radio-frequency microneedles (RF-MN)
- Non-ablative Thulium laser (Active Comparator): Non-ablative Thulium laser (NAFL) single treatment
  Interventions: Device: Non-ablative Thulium laser (NAFL)
- RF microneedles (Active Comparator): Radio-frequency microneedles (RF-MN) single treatment
  Interventions: Device: Radio-frequency microneedles (RF-MN)
- Control (No Intervention): Control receiving no intervention

INTERVENTIONS:
Combination Product: Photodynamic therapy — Photodynamic therapy with Methyl Aminolevulinate creme and red light.
  Arms: RF microneedles + photodynamic therapy; Thulium laser + photodynamic therapy
Device: Non-ablative Thulium laser (NAFL) — Non-ablative Thulium laser (NAFL).
  Arms: Non-ablative Thulium laser; Thulium laser + photodynamic therapy
Device: Radio-frequency microneedles (RF-MN) — Radio-frequency microneedles (RF-MN).
  Arms: RF microneedles; RF microneedles + photodynamic therapy

SUMMARY:
This study investigates a non-ablative fractional thulium laser and a radio-frequency microneedling device as pre-treatment for combination photodynamic therapy in treatment of photoaged skin and actinic keratoses.

DETAILED DESCRIPTION:
Photoaging of skin and actinic keratoses Photoaging of the skin is the result of UV radiation in chronic sun exposure and its deleterious effects. Photoaging includes fine and coarse wrinkles, roughness, laxity, mottled pigmentation, coarseness, sallowness, telangiectasia, solar lentigines and dysplastic actinic keratoses. The process can be of both cosmetic and medical importance. Actinic keratoses (AK) are common dysplastic pre-malignant lesions that may develop into a malign invasive squamous cell carcinomas (SCC). SCCs have metastatic potential at up to 3%. The risk of malign transformation from AK to SCC is highest in chronic sun-damaged skin with confluent field-cancerization from multiple AK. National guidelines recommend treatment of the entire field of sun damaged skin with photodynamic therapy and several topical drugs, e.g. imiquimod, diclofenac, ingenol mebutate, and 5-fluoruracil. Repeat treatments are usually necessary to achieve the desired results in patients with chronic sun damaged skin.

Photochemical treatment with photodynamic therapy

Photodynamic therapy (PDT) is a treatment that uses a photosensitizer drug activated in the skin by light in the visible spectrum. Methyl aminolevulinate (MAL) is a photosensitizing agent with great affinity for dysplastic cells, and transforms into the light-sensitive Protoporphyrin PpIX. When exposed to light, photoactivated PpIX catalyzes a reactive oxygen species reaction, which leads to irreversible cell apoptosis of the dysplastic or neoplastic tissue. PDT can be used as treatment of a wide range of photoaging skin defects including actinic keratoses, and is exceedingly well suited for treatment of larger skin areas. PDT produces cosmetically pleasing results in extension of the excellent AK clearance.

Physical intervention with fractional laser and light-based interventions

Fractional laser and light-based treatments with lasers and microneedles are approaches that can be applied very precisely, and can be used to rejuvenate photodamaged skin.

Laser-treatment for rejuvenation of skin can be achieved using a non-ablative 1927 nm fractionated thulium laser (NAFL), good results have been reported for many aspects of photoaging, and specifically for actinic keratoses with good results. The thulium laser works by creating vertical thermal laser-channels in the skin without the ablative effect to the epidermis. Laser-treatment with the thulium laser may be combined with other treatments like PDT to produce synergistic effects.

Microneedling (MN) is a treatment option in which the skin epidermis is penetrated by closely arranged multiple microneedles. This can induce collagen production and stimulate the release of growth factors, and collagen synthesis and remodeling, producing the effects of rejuvenation. Radio-frequency (RF) microneedling (MN), also known as RF-MN, adds RF making it possible for insulated needles to emit heat at the needle-heads when the epidermis is fully punctured, possibly enhancing the described effects even further. Good results have been reported using MN as skin rejuvenation, and can the treatment be used in conjunction with PDT.

The delicate skin of the décolleté is subject to a high amount of accumulated life-time sun exposure, and is thus highly susceptible to photoaging effects. A mild and effective treatment of photodamaged skin for this particular area is highly desirable, and may be achieved by developing new combination strategies, in which the thulium laser or a microneedling device can be used as effective pre-treatment for PDT. To our knowledge, no previous randomized study has compared the use of the non-ablative thulium laser or microneedling in combination with photodynamic treatment (PDT).

ELIGIBILITY:
Inclusion Criteria:

* Décolleté with chronic field-change photodamaged skin.
* Area with visually homogenous photodamage.
* Provide informed written consent.
* Fertile women must provide a negative U-hCG pregnancy test at the time of inclusion, and use safe anticontraceptive during the entire study period, e.g. oral hormonal contraceptives, intrauterine devices, subdermal implantation, or hormonal vaginal ring.

Exclusion Criteria:

* Treatment of actinic keratoses in the décolleté area within the last 30 days.
* Porphyria.
* Pregnant or nursing women.
* Skin cancer (invasive, in situ), keratoacanthoma, or other infiltrating tumors in the study area.
* Known tendencies to produce hypertrophic scarring or keloids.
* Allergies against Metvix creme solution, peanuts, or soy.
* Considered unable to follow the study protocol, e.g. alcohol dependence syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of photodamage | 12 weeks
  5-point categorial scale of photodamage severity, measuring changes in skin texture, pigmentation, telangiectasia, and wrinkles. Scores are 0, 1, 2, 3, and 4, for none, mild, moderate, severe, and very severe, respectively. A reduction in score from initial scoring to post-treatment is desirable.

SECONDARY OUTCOMES:
Treatment effect on actinic keratoses | 12 weeks
  Evaluated on the Olsen grading scale for actinic keratoses thickness. Scores are 1, 2, and 3, for slightly palpable, moderately thick, and very thick and hyperkeratotic, respectively. A reduction in score from initial scoring to post-treatment is desirable.
Severity of local skin reactions | 7 days
  Local skin reaction (LSR)-grading scale. Evaluation of redness, scaling, edema, pustules, and erosion on a 5-point categorial scale of severity. Scores are 0, 1, 2, 3, and 4, for individual parameters:
  Redness: None, slightly pink <50%, pink or light red >50%, red restricted to treatment area, and red extending outside treatment area.
  Scaling: None, isolated scale, scaling <50%, scaling >50%, scaling extending outside treatment area.
  Edema: None, slight specific edema, palpable edema beyond individual lesions, confluent and/or visible edema, and marked swelling extending outside treatment area.
  Pustules: None, vesicles only, transudate or pustules <50%, transudate or pustules >50%, and transudate or pustules extending outside treatment area.
  Erosion: None, lesion specific erosion, erosion extending beyond individual lesion, erosion >50%, and black eschar or ulceration.
Presence of perceived pain during treatment | 0 days
  VAS Visual analogue scale for perceived pain. Scores are 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10, ranging from none to very severe. Higher is worse, and lower scores for treatment modalities are desirable.
Cosmetic results | 12 weeks
  Cosmetic results on a 5-point categorial scale for perceived cosmetic outcome compared with base starting point for the individual patient. Scores are 0, 1, 2, 3, and 4, for poor, acceptable, good, excellent, and outstanding, respectively. A higher score is desirable.
Protoporphyrin IX (PpIX) fluorescence uptake | 0 days
  Levels of PpIX uptake in the skin computed quantitatively from PpIX imaging. Imaging before application, after 3 hours, and after LED exposure.
Safety including wounding, scarring, hyper and hypo pigmentation | 12 weeks
  Safety concerning side-effects evaluated on a 5-point categorial scale for hyper- and hypopigmentation, erosions, and scarring. Scores are 0, 1, 2, 3, and 4, for none, mild, moderate, severe, and very severe. A lower score is desirable.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No